CLINICAL TRIAL: NCT02229136
Title: Evaluation of Miracle Mouthwash (MMW) Plus Hydrocortisone and Prednisolone Mouth Rinse as Prophylaxis for Everolimus-Associated Stomatitis
Brief Title: Miracle Mouthwash Plus Hydrocortisone vs Prednisolone Mouth Rinse for Mouth Sores Caused by Everolimus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13026; CRAD001JUS240T (Other: Novartis)
Record Dates: First submitted 2014-08-26; First posted 2014-08-29 (Estimated); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Stomatitis; Oral Mucositis; Neoplasm of the Breast; Malignant Tumor of Breast
Keywords: Mouth sores from chemotherapy; mouth sores; hormone receptor-positive metastatic breast cancer; metastatic breast cancer
MeSH Terms: conditions — Stomatitis; Breast Neoplasms; Oral Ulcer | interventions — Hydrocortisone; Prednisolone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Miracle Mouthwash plus Hydrocortisone (Experimental): Miracle Mouthwash plus Hydrocortisone, swish and expectorate 10cc (10 mLs) 4 times per day, every day for 12 weeks.
  Interventions: Drug: Miracle Mouthwash Plus Hydrocortisone
- Prednisolone (Active Comparator): Prednisolone oral solution 15 mg/5 ml; swish and expectorate 10cc (10 mL) 4 times per day, every day for 12 weeks.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Miracle Mouthwash Plus Hydrocortisone — Miracle Mouthwash Plus Hydrocortisone (16 oz recipe/480 ml)
  Arms: Miracle Mouthwash plus Hydrocortisone
Drug: Prednisolone — Prednisolone oral solution 15 mg/5 ml
  Other Names: Millipred; Omnipred; Orapred; Econopred; Flo-Pred
  Arms: Prednisolone

SUMMARY:
This is a randomized Phase 2 study to evaluate two different steroid-based mouth rinses (Miracle Mouth Wash plus hydrocortisone versus prednisolone oral rinse) for the prevention or treatment of everolimus-associated stomatitis (mouth sores) in postmenopausal patients undergoing treatment with an aromatase inhibitor plus everolimus. An exploratory analysis will also evaluate patient response to next anti-cancer therapy of physician's choice following discontinuation of therapy with an aromatase inhibitor plus everolimus.

DETAILED DESCRIPTION:
Stomatitis, or inflammation of the mucous membranes lining the mouth and throat, is a common side affect associated with chemotherapy and radiation therapy. In addition, stomatitis has been reported in approximately 44% - 64% of patients treated with everolimus (Afinitor PI). However, mTOR (mammalian target of rapamycin) inhibitor-induced stomatitis (mIAS) is a different clinical entity, manifesting more frequently as discrete aphthous-like lesions rather than diffuse inflammation. Oral lesions are typically well demarcated, single or multiple ovoid-shaped ulcerations, with a grayish-white pseudomembrane.

In the BOLERO-2 trial, 56% of patients with MBC (metastatic breast cancer) treated with exemestane plus everolimus developed stomatitis, with 37% developing grade 2/3 stomatitis. These rates are consistent with the rates reported with everolimus therapy in patients with other types of cancers (Afinitor PI). Although this adverse event is reversible, approximately one-fourth of the patients treated with everolimus in the BOLERO-2 trial required dose interruptions or dose reductions, and this may impact the benefit from therapy. Despite the frequency of stomatitis associated with mTOR inhibitor therapy, strategies to prevent and/or ameliorate this painful side effect are not well defined or documented. Expert guidelines on the management of mIAS have been developed, but these guidelines are based on retrospective observational and/or anecdotal evidence, and prospective data on the efficacy of mIAS prevention and management strategies are needed.

There is some evidence to suggest steroid therapy may be helpful in the management of mIAS. Steroid-containing ointments or mouth rises have also been shown to alleviate symptoms in patients with non-chemotherapy associated apthous oral ulcers. Reports on the effectiveness of non-steroid mouthwash formulations have been mixed, but agents that induce a topical anesthetic effect, may help to reduce discomfort and pain.

Thus, the present study has been designed to investigate the effectiveness of two oral rinses (miracle mouth wash [MMW] plus hydrocortisone, vs prednisolone) to prevent or reduce the severity of stomatitis in patients with MBC undergoing treatment with an aromatase inhibitor plus everolimus (AIE).

In addition, because very little is known about the impact of everolimus therapy on response to later lines of treatment for MBC, and preclinical data suggest mTOR inhibition may resensitize cells to endocrine therapy, this study will also assess tumor response to next anti-cancer therapy of physician's choice, including duration of response and sites of progression.

All patients will receive everolimus 10 mg PO QD (by mouth, every day) plus standard dose AI (physician choice of Letrozole, Exemestane, or Anastrozole).

Patients will be randomized 1:1 to 12 weeks of treatment with either:

* Arm 1: MMW plus hydrocortisone
* Arm 2: Prednisolone oral solution (15mg/5ml)

Treatment with the oral rinse will start on Day 1 of everolimus therapy, and will be self-administered. Patients will be instructed to swish and expectorate (cough or spit out) 10ml of the assigned mouth rinse 4 times per day. Patients may also gargle 4 times per day with the assigned rinse for any symptoms of pharyngitis. Patients will also be instructed to fill out the Oral Stomatitis Daily Questionnaire (OSDQ) at home every day.

The incidence of stomatitis, as well as other adverse events, dose reductions/interruptions, and everolimus discontinuation due to toxicity, will be monitored for the first 12 weeks of treatment. After the end of the initial 12 week randomized portion of the study, patients will continue to be followed every 2 months (for up to 1 year following discontinuation of everolimus for progression or intolerable toxicity or progression on subsequent anti-cancer therapy, whichever occurs first) to determine when AIE treatment is discontinued and reason for discontinuation (toxicity, progression), sites of disease progression, response to next anti-cancer therapy of physician's choice (by physician assessment) and duration of response, and sites of disease progression to next anti-cancer therapy following progression on AIE.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. ECOG (Eastern Cooperative Group) Performance status ≤ 2;
3. Histologic or cytologic confirmation of stage IV hormone receptor-positive breast cancer;
4. Postmenopausal status, defined either by:

   1. Age ≥ 55 years and ≥ 1 year of amenorrhea
   2. Age < 55 years and ≥ 1 year of amenorrhea, with an estradiol assay <20pg/ml
   3. Surgical menopause with bilateral oophorectomy Note: Ovarian radiation or treatment with a luteinizing hormone-releasing hormone (LHRH) agonist (goserelin acetate or leuprolide acetate) is not permitted for induction of ovarian suppression;
5. Planned treatment with an aromatase inhibitor (letrozole, exemestane, or anastrozole) plus everolimus; Note: Prior treatment with an aromatase inhibitor, either for early-stage or metastatic breast cancer, is allowed.
6. Adequate bone marrow function as shown by: ANC (absolute neutrophil count) ≥1.5 x 109/L, Platelets ≥100 x 109/L, Hb >9 g/dL;
7. Adequate liver function as shown by:

   1. Total serum bilirubin ≤2.0 mg/dL,
   2. ALT (Alanine aminotransferase) and AST (Aspartate aminotransferase) ≤2.5x ULN (upper limit of normal) (≤5x ULN in patients with liver metastases),
   3. INR (International Normalized Ratio) ≤2;
8. Adequate renal function: serum creatinine ≤1.5x ULN;
9. Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤2.5x ULN.

   Note: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication;
10. Willingness to complete a daily stomatitis symptom questionnaire;
11. Signed informed consent obtained prior to any screening procedures.

Exclusion Criteria:

1. Known intolerance or hypersensitivity to everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus);
2. Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral everolimus;
3. Uncontrolled diabetes mellitus as defined by HbA1c (hemoglobin A1c) >8% despite adequate therapy. Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary;
4. Patient has any severe and/or uncontrolled medical conditions such as:

   1. unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to start of Everolimus, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease
   2. Symptomatic congestive heart failure of New York Heart Association Class III or IV
   3. active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and chronic hepatitis (i.e. quantifiable HBV-DNA (Hepatitis B Virus DNA) and/or positive HbsAg, quantifiable HCV-RNA [Hepatitis C Virus RNA]),
   4. known severely impaired lung function (spirometry and DLCO [Diffusing capacity of the Lung for Carbon Monoxide] 50% or less of normal and O2 saturation 88% or less at rest on room air),
   5. active, bleeding diathesis;
5. Patient requires chronic treatment with corticosteroids (including inhaled corticosteroids) or other immunosuppressive agents. Topical corticosteroids are allowed;
6. Known history of HIV seropositivity;
7. Patient received live attenuated vaccines within 1 week of start of everolimus and during the study. Patient should also avoid close contact with others who have received live attenuated vaccines. Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG (Bacillus Calmette-Guérin), yellow fever, varicella and TY21a typhoid vaccines;
8. Patient has a history of another primary malignancy, with the exceptions of: non-melanoma skin cancer, and carcinoma in situ of the cervix, uteri, or breast from which the patient has been disease free for ≥3 years;
9. Patient has a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study;
10. Patient is currently part of or has participated in any clinical investigation with an investigational drug within 1 month prior to dosing.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Grade ≥ 2 stomatitis | 12 weeks
  The primary objective of the study is to determine the incidence of Grade ≥ 2 stomatitis in patients undergoing treatment with an aromatase inhibitor plus everolimus (AIE) when treated with either Miracle Mouthwash (MMW) plus hydrocortisone or with a prednisolone mouth rinse during the first 12 weeks of treatment.

SECONDARY OUTCOMES:
Incidence of all side effects | 64 weeks
  Determination of the incidence of adverse events (all grades)
Percentage of patients requiring dose interruptions and/or dose reductions of everolimus | 64 weeks
  Determination of the percentage of patients requiring dose interruptions and/or dose reductions of everolimus, as well as the percentage of patients discontinuing therapy with everolimus due to toxicity.
Reduction in pain score on questionnaires | 12 weeks
  Evaluation of the impact of MMW plus hydrocortisone or a prednisolone mouth rinse on the duration and severity of stomatitis, as assessed by the Oral Stomatitis Daily Questionnaire (OSDQ).

OTHER OUTCOMES:
Time to Disease Progression of next anti-cancer therapy | 64 weeks
  An exploratory objective is to assess patient response to the next anti-cancer therapy of physician's choice following progression on AIE, including duration of response and sites of progression.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce A. O'Shaughnessy, MD, Principal Investigator — US Oncology Research, McKesson Specialty Health
Locations (1):
- 12 sites incl Yakima, WA, Boulder, CO, and Austin, TX, US, Texas, United States